CLINICAL TRIAL: NCT02219698
Title: Symptomatic Treatment of Acute Uncomplicated Diverticulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Vatsatautien tutkimussäätiö - foundation (Unknown); Mary and Georg Ehrnroot's foundation (Unknown); Finnish Surgical society (Unknown); Martti I. Turunen Foundation (Unknown); Governmental competitive funds (EVO) (Unknown)
Responsible Party: Principal Investigator, Ville Sallinen, M.D., Ph.D., Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS-Dnro122-2014
Record Dates: First submitted 2014-08-11; First posted 2014-08-19 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Ibuprofen; Acetaminophen

ARMS (1):
- Symptomatic treatment (Experimental)
  Interventions: Drug: Ibuprofen; Drug: Paracetamol

INTERVENTIONS:
Drug: Ibuprofen
Drug: Paracetamol

SUMMARY:
The purpose of this study is to determine the safety and efficacy of symptomatic treatment (i.e. without antimicrobial drugs) of acute uncomplicated diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

* Computed tomography-diagnosed acute uncomplicated* diverticulitis

  * No abscess, fistula, obstruction and distant intra- or retroperitoneal air. Pericolic air allowed.

Exclusion Criteria:

* Already commenced antimicrobial medication
* Immunosuppression (e.g. diabetes, corticosteroid medication, immunosuppressive medication, chemotherapy, chronic liver disease)
* Suspicion of generalized peritonitis
* Organ dysfunction
* Another infection requiring antimicrobial medication
* Pregnancy
* Age < 18 years or > 90 years
* Missing written consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Complications of diverticulitis | 30 days from allocation
  Incidence of complications of diverticulitis (abscess, free perforation, need for surgery)

SECONDARY OUTCOMES:
Length of hospital stay (days) | At the end of the hospital stay, an expected average of 2 days
Rate of re-admissions | 30 days from discharge
  Number patients re-admitted to hospital
Recurrence of diverticulitis | 10 years
  Number of recurrent diverticulitis within follow-up
Mortality | 30 days from allocation
  Number of patients deceased
Need for elective sigmoid resection | 10 years
  Number of patients that have undergone elective sigmoid resection
Need for emergency surgery for diverticulitis on another admission | 10 years
  Number of patients requiring emergency surgery for diverticulitis on another admission
Commencement of antimicrobial drug | For the duration of hospital stay, an expected average of 2 days
  Number of patients that have received antimicrobial drugs
Late complication of diverticulitis | 10 years
  Number of patients who develop late complications of diverticulitis e.g. fistula, stricture
Stoma rate | 10 years
  Number of patients who receive a stoma

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Mali JP, Mentula PJ, Leppaniemi AK, Sallinen VJ. Symptomatic Treatment for Uncomplicated Acute Diverticulitis: A Prospective Cohort Study. Dis Colon Rectum. 2016 Jun;59(6):529-34. doi: 10.1097/DCR.0000000000000579. PMID 27145310